CLINICAL TRIAL: NCT02163421
Title: A Phase 1, Open Label, Randomized, Parallel Group Study to Assess the Absolute Bioavailability and Pharmacokinetics of Vedolizumab in Healthy Participants Following Single Subcutaneous Administration
Brief Title: Bioavailability and Pharmacokinetics of Vedolizumab in Healthy Participants Following Single Subcutaneous Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MLN0002SC_101; 2014-000927-26 (EudraCT Number); U1111-1152-6903 (Registry Identifier: WHO); 14/LO/0466 (Registry Identifier: NRES)
Record Dates: First submitted 2014-06-06; First posted 2014-06-13 (Estimated); Results first posted 2017-02-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-12

CONDITIONS: Healthy
Keywords: Drug therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vedolizumab SC 54 mg (Experimental): Vedolizumab SC, once on Day 1.
  Interventions: Drug: Vedolizumab SC
- Vedolizumab SC 108 mg (Experimental): Vedolizumab SC, once on Day 1.
  Interventions: Drug: Vedolizumab SC
- Vedolizumab SC 160 mg (Experimental): Vedolizumab SC, once on Day 1.
  Interventions: Drug: Vedolizumab SC
- Vedolizumab IV 300 mg (Active Comparator): Vedolizumab IV, once on Day 1.
  Interventions: Drug: Vedolizumab IV

INTERVENTIONS:
Drug: Vedolizumab SC — Vedolizumab injection, for subcutaneous use (vedolizumab SC)
  Other Names: MLN0002SC
  Arms: Vedolizumab SC 108 mg; Vedolizumab SC 160 mg; Vedolizumab SC 54 mg
Drug: Vedolizumab IV — Vedolizumab injection, for intravenous use (vedolizumab IV)
  Other Names: MLN0002SC
  Arms: Vedolizumab IV 300 mg

SUMMARY:
The purpose of this study is to assess the absolute bioavailability and pharmacokinetics of vedolizumab following a single injection of vedolizumab subcutaneously at 3 varying doses.

DETAILED DESCRIPTION:
The drug being tested in this study is called vedolizumab. Vedolizumab is being tested to determine its bioavailability, safety, and tolerability in the body with three varying doses of vedolizumab SC compared to people who are administered vedolizumab IV.

The study will enroll approximately 24 non-Japanese patients and 24 Japanese patients. Participants will be randomly assigned to one of the four treatment groups:

* Vedolizumab Intravenous 300 mg
* Vedolizumab Subcutaneous 54 mg
* Vedolizumab Subcutaneous 108 mg
* Vedolizumab Subcutaneous 160 mg

All participants will receive the treatment they are assigned on Day 1 of the study.

This single-center trial will be conducted in the United Kingdom. The overall time to participate in this study is up to 196 days. Participants will make 10 visits to the clinic, including one 8 day period of confinement to the clinic, and will be contacted by telephone at Study Day 168 (+/-3), approximately 6 months after dose for a follow-up questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant, or when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Is a healthy male or female adult of non-Japanese decent 18 to 60 years of age inclusive or of Japanese descent (born to Japanese parents and grandparents and has lived outside Japan for less than 5 years), 20 to 60 years of age inclusive, at the time of informed consent.
4. Weighs at least 45 kg (99 lb) and have a body mass index (BMI) between 18.0 and 30.0 kg/m^2 for non-Japanese participants or 18.0 and 28.0 kg/m^2 for Japanese participants, inclusive at Screening.
5. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for a minimum of 18 weeks after last dose.
6. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use acceptable methods of contraception from signing of informed consent throughout the duration of the study and for a minimum of 18 weeks after last dose.

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to dosing of study medication or history of treatment with another monoclonal antibody within 6 months to dosing of study medication.
2. Has received vedolizumab in a previous clinical study or as a therapeutic agent.
3. Is an immediate family member, study site employee, or in a dependant relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
4. Has uncontrolled, clinically significant (CS) neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, endocrine disease, or psychiatric disorder, or other abnormality, that may impact the ability of the participant or potentially confound the study results.
5. Has a known hypersensitivity to any component of the formulation of vedolizumab SC or vedolizumab IV.
6. Has one or more positive responses on the progressive multifocal leukoencephalitis (PML) subjective symptom checklist at screening or before dosing on Day 1.
7. Has a positive result for drugs of abuse or alcohol at Screening or Check- in (Day -1).
8. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the Screening visit or is unwilling to agree to abstain from alcohol for 48 hrs prior to Day -1 throughout confinement and for 48 hrs prior to each clinic visit and drugs throughout the study.
9. Is pregnant or lactating or intends to become pregnant before, during, or within 18 weeks after the last dose in this study; or intends to donate ova during such time period.
10. If male, the participant intends to donate sperm during the course of this study or for 18 weeks after the last dose in this study.
11. Has evidence of current cardiovascular, central nervous system, hepatic, hematopoietic disease, renal dysfunction, metabolic or endocrine dysfunction, serious allergy, asthma hypoxemia, hypertension, seizures, or allergic skin rash. There is any finding in the participant's medical history, physical examination, or safety laboratory tests giving reasonable suspicion of a disease that would contraindicate taking vedolizumab, or a similar drug in the same class, or that might interfere with the conduct of this study. This includes, but is not limited to, peptic ulcer disease, seizure disorders, and cardiac arrhythmias.
12. Had a surgical procedure requiring general anesthesia within 30 days before the initial Screening Visit, or is planning to undergo a surgery that requires general anesthesia during the study period through Final Visit Day 127.
13. Has a history of cancer, except basal cell carcinoma that has been in remission for at least 5 years prior to Day 1.
14. Participant is unable to attend all study days or comply with protocol requirements.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United Kingdom from 09 June 2014 to 16 January 2015.
Pre-assignment Details: Healthy participants of age group 18 years to 60 years were enrolled in 1 of the 4 treatment groups: Vedolizumab intravenous 300 milligram (mg); Vedolizumab subcutaneous 54 mg; Vedolizumab SC 108 mg and Vedolizumab SC 160 mg.
Groups:
- Vedolizumab Intravenous 300 mg: Vedolizumab 300 mg, 30-minutes infusion, intravenously once only on Day 1 in a treatment period of 168 days.
- Vedolizumab Subcutaneous 54 mg: Vedolizumab 54 mg, injection, subcutaneously, once only on Day 1 in a treatment period of 168 days.
- Vedolizumab Subcutaneous 108 mg: Vedolizumab 108 mg, injection, subcutaneously, once only on Day 1 in a treatment period of 168 days.
- Vedolizumab Subcutaneous 160 mg: Vedolizumab 160 mg, injection, subcutaneously, once only on Day 1 in a treatment period of 168 days.
Period: Overall Study
Arm/Group | Vedolizumab Intravenous 300 mg | Vedolizumab Subcutaneous 54 mg | Vedolizumab Subcutaneous 108 mg | Vedolizumab Subcutaneous 160 mg
Started | 12 | 12 | 12 | 12
Completed | 12 | 12 | 12 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all randomized participants who received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vedolizumab Intravenous 300 mg | Vedolizumab Subcutaneous 54 mg | Vedolizumab Subcutaneous 108 mg | Vedolizumab Subcutaneous 160 mg | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (12.30) | 41.0 (13.06) | 31.1 (9.59) | 35.2 (12.89) | 35.3 (12.21)
Gender [Count of Participants; unit: Participants]
  Female | 4 | 5 | 5 | 5 | 19
  Male | 8 | 7 | 7 | 7 | 29
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 6 | 6 | 6 | 6 | 24
  White | 5 | 6 | 6 | 6 | 23
  Multiracial | 1 | 0 | 0 | 0 | 1
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 65.8 (13.84) | 68.0 (12.96) | 67.6 (13.42) | 64.3 (14.58) | 66.4 (13.35)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 21.8 (2.90) | 23.0 (2.98) | 22.8 (2.44) | 22.0 (3.41) | 22.4 (2.90)
Smoking Classification [Number; unit: participants]
  Had Never Smoked | 8 | 9 | 10 | 6 | 33
  Current Smoker | 3 | 1 | 2 | 5 | 11
  Ex-Smoker | 1 | 2 | 0 | 1 | 4
Alcohol Classification [Number; unit: participants]
  Had Never Drunk | 0 | 0 | 1 | 1 | 2
  Current Drinker | 11 | 9 | 9 | 9 | 38
  Ex-Drinker | 1 | 3 | 2 | 2 | 8
Female Reproductive Status [Number; unit: participants] — Female reproductive status was classified as postmenopausal female and female of childbearing potential. None of the female was reported as surgically sterile.
  participants
    Postmenopausal Female | 0 | 1 | 0 | 0 | 1
    Female of Childbearing Potential | 4 | 4 | 5 | 5 | 18
    Not Applicable (Participant was Male) | 8 | 7 | 7 | 7 | 29

OUTCOME MEASURES:

1. Primary Outcome: Population Mean Estimate for Bioavailability Following Subcutaneous (SC) Administration
Description: Bioavailability is defined as the rate and extent to which the active moiety of the e.g. subcutaneous administered drug reaches the systemic circulation. Population mean estimate for bioavailability was based on population pharmacokinetic (PK) analysis to find one measure. The exposure data were pooled across visits and subjects to identify population PK parameter estimates and covariate effects. The outcome measure data was planned to be analyzed using a model collating all arms measures to report pooled data across arms, as per planned analysis. Bioavailability was estimated using population pharmacokinetic (popPK) analysis.
Time Frame: Day 1: predose and on multiple time points (up to Day 127)
Population: The pharmacokinetic analysis set included all randomized participants who received study treatment and who had at least 1 measurable pharmacokinetic concentration.
Measure: Number (95% Confidence Interval); unit: percentage of drug
Groups:
- Vedolizumab Subcutaneous: Vedolizumab 54 mg or 108 mg or 160 mg, injection, subcutaneously, once only on Day 1 in a treatment period of 168 days.
Arm/Group | Vedolizumab Subcutaneous
Number analyzed (Participants) | 36
percentage of drug | 0.751 [0.689 to 0.819]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 168 days after the last dose of study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Vedolizumab Intravenous 300 mg | Vedolizumab Subcutaneous 54 mg | Vedolizumab Subcutaneous 108 mg | Vedolizumab Subcutaneous 160 mg
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 9/12 | 8/12 | 11/12 | 8/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vedolizumab Intravenous 300 mg (N=12) | Vedolizumab Subcutaneous 54 mg (N=12) | Vedolizumab Subcutaneous 108 mg (N=12) | Vedolizumab Subcutaneous 160 mg (N=12)
Headache (Nervous system disorders) | 3 | 3 | 3 | 0
Presyncope (Nervous system disorders) | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 1 | 0
Vessel puncture site swelling (General disorders) | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 1 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 2 | 2 | 3
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 1 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.